CLINICAL TRIAL: NCT01490112
Title: Regulatory Post Marketing Surveillance Study of NovoRapid for New Drug Re-examination
Brief Title: Surveillance Study of NovoRapid® for New Drug Re-examination
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ANA-1881
Record Dates: First submitted 2011-12-06; First posted 2011-12-12 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IAsp
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: insulin aspart — Subjects who had a first drug date on NovoRapid® were prescribed to inject insulin aspart using vial, FlexPen, NovoLet or Penfill devices. Injected subcutaneously (s.c., under the skin) immediately before meals for 24 weeks

SUMMARY:
This study is conducted in Asia. The aim of this study is to observe the safety and efficacy of insulin aspart (NovoRapid®) administered via vial and three different devices.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diabetes mellitus (type 1, type 2, or gestational) prescribed with insulin aspart (NovoRapid®)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with diabetes mellitus (type 1, type 2, or gestational) prescribed with insulin aspart (NovoRapid®)
Sampling Method: Non-Probability Sample
Enrollment: 1239 (Actual)
Dates: Start 2005-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change in weight

SECONDARY OUTCOMES:
Fasting blood glucose (FBG)
HbA1c (glycosylated haemoglobin)
Adverse events: Serious and non-serious

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Seoul, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com